CLINICAL TRIAL: NCT03604133
Title: Ambulatory Surgical Center Implantable Cardioverter-Defibrillator Outcomes Registry
Acronym: ASC ICD Reg
Status: Recruiting | Type: Observational
Sponsor: QuesGen Systems Inc (Other)
Collaborators: Cardio Surgical Partners (Network)
Responsible Party: Sponsor
Other Study IDs: 2018-310 Cardiac Registry
Record Dates: First submitted 2018-07-18; First posted 2018-07-27 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients receiving ICD devices

SUMMARY:
The primary objectives for the registry is to evaluate the overall incidence of serious complications or adverse events for primary implants and replacement devices, and assess the cost and time efficiency for both physicians and patients. The Registry is a multi ASC data collection registry. Data collection will occur at the time of screening, implant, and 2 weeks after implant at the time of wound check.

ELIGIBILITY:
Inclusion Criteria:

* Physician recommendation to receive the implant in an Ambulatory Surgical Center (ASC)

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals who require ICD to maintain optimal health.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-08-24 (Actual); Primary Completion 2023-08-24 (Estimated); Study Completion 2028-08-24 (Estimated)

PRIMARY OUTCOMES:
Successful Implantation | Two-week follow-up assessment
  Patient undergoes surgery for ICD device implantation

CONTACTS AND LOCATIONS:
Locations (1):
- Cardio Surgical Partners, LLC, Lehi, Utah, United States